CLINICAL TRIAL: NCT05226143
Title: A Single Center, Clinical Study to Determine the Safety and Efficacy of an Eczema Spot Treatment in Providing Eczema Symptoms Relief and Lasting Itch Relief to Affected Skin Area
Brief Title: A Study of an Eczema Spot Treatment in Providing Eczema Symptoms Relief and Lasting Itch Relief to Affected Skin Area
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johnson & Johnson Consumer Inc. (J&JCI) (Industry)
Responsible Party: Sponsor
Organization: Johnson & Johnson Consumer and Personal Products Worldwide (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CCSSKA004706
Record Dates: First submitted 2022-01-26; First posted 2022-02-07 (Actual); Last update posted 2022-11-14 (Actual); Status verified 2022-11

CONDITIONS: Dermatitis, Atopic
Keywords: Itching; Pruritus; Dryness; Excoriation; Xerosis; Eczema; Atopic Dermatitis
MeSH Terms: conditions — Dermatitis, Atopic; Pruritus; Eczema

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Gel Cream (Experimental): Participants will be provided with the Gel Cream to apply on clean, dry face (facial skin) once per day and on the target lesion on the face or body at least 2 times per day or more as needed, in the morning and at night for 14 days.
  Interventions: Other: Gel Cream

INTERVENTIONS:
Other: Gel Cream — Gel Cream
  Other Names: Participants will apply gel cream on facial skin and target lesions for up to 14 days.

SUMMARY:
The purpose of this study is to evaluate the efficacy (assessed by clinical evaluation of eczema/atopic lesion severity [atopic dermatitis severity index {ADSI} scoring] and perceived benefits in itch [visual analog score {VAS} scoring]) and tolerability (assessed by clinical grading) of an investigational spot treatment Gel Cream when used on a target site of participants with mild to moderate atopic dermatitis.

ELIGIBILITY:
Inclusion Criteria:

* Fitzpatrick Skin Type I, II, III, IV, V, or VI
* Self-reported natural skin tone Pale/fair to light white, White to light beige, Beige to light tan/light olive, Medium tan/medium olive to light brown, Medium brown to dark brown, or Darkest brown to darkest black targeting the following: a) Skin tones "Pale/fair to light white" and "White to light beige" (at least number of participants (n)= 4); b) Skin tones "Beige to light tan/light olive" and "Medium tan/medium olive to light brown" (at least n = 4); c) Skin tones "Medium brown to dark brown" and "Darkest brown to darkest black" (at least n = 4)
* Men who are regular shavers (at least 3 times per week) and do not have beards. A mustache and/or small goatee is allowed as long as the majority of the face and neck are shaved
* Has mild to moderate eczema severity rating at Visit 1, defined as a score of 3 - 7.5 on the Rajka and Langeland Severity Index
* Has at least 1 lesion area; either on face or body at Visit 1 with a score of 5 - 12 on the Atopic Dermatitis Severity Index (ADSI) score, ADSI pruritus sub-score of 1 - 2 (mild - moderate), and ADSI erythema sub-score of at least 2 (moderate) to be followed for the duration of the study
* Has a Visual Analog Score (VAS) score greater than or equal to (>=) 4 for itch on the target lesion
* Has experienced a recent (within the past 1 year) itch flare up and is currently experiencing preflare up symptoms at Visit 1
* Is a regular user of body moisturizers, defined as 2 -3 times per week
* Has not had any facial treatments in the past 6 months and is willing to withhold all facial treatments during the course of the study including facials, facial peels, photo facials, laser treatments, dermabrasion, botulinum toxin (Botox), injectable filler treatments, intense pulsed light (IPL), acid treatments, tightening treatments, facial plastic surgery, or any other treatment administered by a physician or skin care professional designed to improve the appearance or firmness of facial skin
* Generally in good health based on medical history reported by the participant
* Able to read, write, speak, and understand English
* Individual has signed the Consent for Photograph Release and informed consent document (ICD) including Health Insurance Portability and Accountability Act (HIPAA) disclosure
* Intends to complete the study and is willing and able to follow all study instructions

Exclusion Criteria:

* Has known allergies or adverse reactions to common topical skincare products or ingredients in the investigational study material (ISM)
* Presents with a health condition and/or pre-existing acute or chronic dermatologic conditions (example, psoriasis, rosacea, rashes, many and/or severe excoriations, Et cetera [etc.]) that could interfere with the outcome of the study or be deemed inappropriate for study participation as determined by the principal investigator (PI)
* Has severe eczema severity rating at Visit 1, defined as a score of 8 - 9 on the Rajka and Langeland Severity Index
* Has a bacterial, fungal, or viral skin infection or is susceptible to cutaneous infections
* Is currently using an over-the-counter (OTC) moisturizer specifically indicated for eczema (Active Ingredient: 1 percent [%] - 2% Colloidal Oatmeal stated in the Drug Facts Box) within 3 days prior to Visit 1
* Is currently using Class I-III topical corticosteroids or systemic medications that will affect or have an indirect effect on his/her eczema (including but not limited to betamethasone, clobetasol, desoximetasone, diflorasone, fluocinonide, fluticasone, halcinonide, halobetasol, and mometasone) or have used the aforementioned medications within 4 weeks before study enrollment. (participants on a stabilized regimen of antihistamines for allergy are permitted into the study)
* Has a history of immunosuppression/immune deficiency disorders (including human immunodeficiency virus [HIV] infection or acquired immunodeficiency syndrome [AIDS]) or currently using immunosuppressive medications (example, azathioprine, belimumab, cyclophosphamide, Enbrel, Imuran, Humira, mycophenolate mofetil, methotrexate, prednisone, Remicade, Stelara.), and/or radiotherapy
* Has used an over-the-counter (OTC) hydrocortisone/steroid and/or prescribed topical medications within 2 weeks prior to Visit 1
* Has used an OTC anti-itch spot treatment within 1 week prior to Visit 1
* Has applied moisturizers on the face and/or body within 3 days prior to Visit 1
* Has a history of a confirmed or suspected COVID-19 infection within 30 days prior to the study visit.
* Within 14 days prior to Visit 1, has been in close contact (exposure within 6 feet for a cumulative time of 15 minutes or more over a 24-hour period) with anyone who has been infected with COVID-19
* Is under a COVID-19 isolation/quarantine order
* Has experienced any of the following self-reported symptoms of COVID-19 within 2 weeks prior to the study visit: a) Unexplained cough, shortness of breath/difficulty breathing, fatigue, body aches (headaches, muscle pain, stomachaches), conjunctivitis, loss of smell, loss of taste, poor appetite, nausea, vomiting, diarrhea, palpitations, or chest pain/tightness; b) Temperature greater than or equal to (>=) 37.2 degree Celsius (°C) / 99 degree Fahrenheit (°F), measured; c) Use of fever or pain reducers within 2 days prior to the study visit
* Has self-reported Type 1 or Type 2 diabetes or is taking insulin or another anti-diabetic medication
* Is taking a medication that would mask an Adverse Event (AE) or confound the study results, including: a) Prescription medication (oral or topical) that can make skin more sensitive or have an effect on the skin (that is, antibiotics, hormones, insulin, etc.) within 6 weeks before Visit 1; b) Immunosuppressive or steroidal drugs within 2 months before Visit 1; c) Non-steroidal anti-inflammatory drugs within 5 days before Visit 1; d) Antihistamines within 2 weeks before Visit 1
* Is self-reported to be breastfeeding, pregnant or planning to become pregnant during the study
* Has a history of or a concurrent health/other condition/situation which may put the individual at significant risk, confound the study results, or interfere significantly with the individual's participation in the study
* Has started prescription testosterone therapy less than 3 months prior to study entry or planning on starting, stopping, or changing doses of testosterone therapy during the study (example, testosterone cypionate, testosterone enanthate, testosterone pellet, testosterone undecanoate) or on a testosterone booster or prescription testosterone (example, DHEA, Omnadren, Sustanon, testosterone cypionate, testosterone enanthate, testosterone propionate, testosterone phenylpropionate, tribulus)
* Has planned surgeries and/or invasive medical procedures during the course of the study
* Is simultaneously participating in any other clinical study or has participated in any product-use study within 30 days prior to Visit 1
* Is an employee/contractor or immediate family member of the PI, Study Site, or Sponsor

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2022-02-21 (Actual); Primary Completion 2022-03-09 (Actual); Study Completion 2022-03-09 (Actual)

PRIMARY OUTCOMES:
Rajka and Langeland Severity Index Score of Target Lesion | At Screening
  Rajka and langeland severity index score of target lesion will be reported. The score is based on the grading of: (i) eczema extent based on percent (%) body area affected, (ii) eczema course based on the number of months with remission during the previous year, and (iii) eczema intensity expressed in terms of nocturnal sleep disturbance due to itch. Each parameter is scored on a scale of 1-3, and the scores are summed. The Rajka and Langeland severity score ranges from 3 to 9 (3-4=mild, 4.5-7.5=moderate, and 8-9=severe).
Atopic Dermatitis Severity Index (ADSI) Score of Target Lesion | Up to 14 days
  ADSI score of target lesion will be reported. ADSI is a scoring system that reflects the severity of a target eczema lesion. The ADSI score is a sum of scores for 5 different parameters - erythema, pruritus, exudation, excoriation, lichenification- which are each measured on a scale of 0 (none) to 3 (severe). The total score can range from 0 (no eczema signs) to 15 (severe eczema lesion).
Dryness of Target Lesion | Up to 14 days
  Dryness of target lesion will be reported. It will be evaluated on a scale of 0 to 3 with 0=none (no dryness), 1=mild (slight, but definite dryness), 2=moderate (definite dryness), and 3=severe (marked dryness), with higher scores indicating a worse outcome.
Tactile Roughness of Target Lesion | Up to 14 days
  Tactile roughness of target lesion will be reported. It will be evaluated on a scale of 0 to 3 with 0=none (skin perfectly smooth), 1=mild (mild roughness), 2=moderate (moderate roughness), and 3=severe (severe roughness), with higher scores indicating a worse outcome.
Erythema of Target Lesion | Up to 14 days
  Erythema of target lesion (derived from ADSI sub-score) will be reported. It will be evaluated on a scale of 0 to 3 with 0=none (no redness), 1=mild (mildly detectable erythema; pink), 2=moderate (dull red; clearly distinguishable), and 3=severe (deep, dark red; marked and extensive), with higher scores indicating a worse outcome.
Pruritus of Target Lesion | Up to 14 days
  Pruritus of target lesion (derived from ADSI sub-score) will be reported. It will be evaluated on a scale of 0 to 3 with 0=none (no itching), 1=mild (occasional, slight itching), 2=moderate (frequent or intermittent itching; does not disturb sleep), and 3=severe (constant, bothersome itching that disturbs sleep or normal activity), with higher scores indicating a worse outcome.
Skin Tone of Lesion Compared to Normal Overall Skin Tone | Up to 14 days
  Skin tone of lesion compared to normal overall skin tone will be reported. It will be evaluated on a scale of 0 to 9 with 0=none (same overall tone [color] of normal, non-involved lesional skin), 1-3=mild (slightly different color/skin tone compared to normal, non-involved lesional skin), 4-6=moderate (moderately different color/skin tone compared to normal, non-involved lesional skin), and 7-9=severe (marked, severe difference in color/skin tone [either hypo/hyper pigmented, red] compared to normal, non-involved lesional skin), with higher scores indicating a worse outcome.
Overall Irritation of Facial Skin | Up to 14 days
  Overall irritation of the facial skin will be reported. It will be evaluated on a scale of 0 to 4 with 0=none (no Reaction), 1=mild (definite pink to red coloration), 2=moderate (increased redness, possible edema), 3=severe (very red, with edema and vesiculation), 4=very severe (deep red, swelling and edema with signs of bullae formation and necrosis), with higher scores indicating a worse outcome.
Itch Assessment of Target Lesion | Up to 14 days
  Itch assessment of target lesion will be evaluated by using visual analog scale (VAS). Participants will be asked to rate his/her itch severity of the target lesion using VAS as score ranges from 0 (no itch) to 10 (worst itch possible).
Soothing Assessments of Target Lesion | Up to 14 days
  Soothing assessment based on participants self-assessment questionnaire score will be reported. Participants will be asked to complete the following question: 1) the product soothed/calmed the eczema test site area; 2) the eczema test site area feels soothed/calmed. Participant responses for each question will have 5 response options such as: Strongly agree, Agree, Neither Agree nor Disagree, Disagree, Strongly Disagree.
Cooling Assessment of Target Lesion | Baseline (Day 0)
  Cooling assessment of target lesion based on participants self-assessment questionnaire score will be reported. Participants will be asked to complete the following question: "The product provided a cooling sensation to the test site area". Participant responses for the question will have 5 response options such as: Strongly agree, Agree, Neither Agree nor Disagree, Disagree, Strongly Disagree.
Burning/Stinging Sensation of the Facial Skin | Up to 14 days
  Burning/Stinging sensation of the facial skin will be reported. It will be evaluated on a scale of 0 to 3 with 0=none (no burning/stinging of the treatment area), 1=mild (slight burning/stinging sensation of the treatment area; slightly bothersome), 2=moderate (definite burning/stinging of the treatment area that is somewhat bothersome), and 3=severe (intense burning/stinging sensation of the treatment area that causes definite discomfort and may interrupt daily activities and/or sleep), with higher scores indicating a worse outcome.
Skin pH Measurements of Target Lesion | Up to 14 days
  Skin pH measurement of target lesion will be reported. It will be measured using a DermaLab pH probe attached to a Cortex Technologies computer platform.
Skin Hydration of Target Lesion as Measured by Corneometer | Up to 14 days
  Skin hydration of target lesion as measured by Corneometer will be reported. Corneometer measurements will be taken using a DermaLab pin probe attached to a Cortex Technologies computer platform.
Transepidermal Water Loss (TEWL) Measurement of Target Lesion | Up to 14 days
  TEWL measurement of target lesion will be assessed. TEWL measurements will be taken using a RG-1 Evaporimeter (cyberDERM) equipped with DermaLab (Cortex Technologies) probes in conjunction with a computer.
Digital Photograph of Target Lesion | Up to 14 days
  Digital photograph of target tension will be reported. The images of each participant's target lesion will be captured using a Canfield D90 digital Slue camera using visible light. This will allow fixed to stop reproducible images to be obtained. A close-up image will be taken of each target lesion with an appropriately draped background.
Microbiome Sampling of Target Lesion | Up to 14 days
  The surface skin microbiome will be collected from target lesion. A swabbing technique will be used to collect surface skin microflora for analysis to determine the effect of the gel cream on the skin microflora.
Itch Quality of Life (ItchQOL) Questionnaire | Up to 14 days
  ItchQOl is a 54-item questionnaire assessing the pruritus-specific disease burden on 2 domains: frequency and bother. The responses to the frequency items are scored on a 1 (never) to 5 (all the time) scale and the responses to the bother items are scored on a 1 (not bothered) to 5 (severely bothered) scale. Higher scores indicate a more adverse impact on quality of life.
Dermatology Life Quality Index (DLQI) Score | Up to 14 days
  The DLQI is a validated questionnaire used to measure the impact of atopic dermatitis (AD) disease symptoms and treatment on health-related quality of life. DLQI consisting of a set of 10 questions which assess quality of life over the past week. Responses to each questions were assessed on a scale of 0 to 3, where 0 is "not at all or not relevant" and 3 is "very much". Scores from all 10 questions added up to give total DLQI scores ranged from 0 (no effect at all on participant's life) to 30 (extremely large effect on participant's life), higher scores indicated more impact on quality of life.
Final Assessment Questionnaire | At Day 14
  Final assessment questionnaire will be completed by the participant to provide subjective assessment of the gel cream. Participant responses for each question will have 5 response options such as: Strongly agree, Agree, Neither Agree nor Disagree, Disagree, Strongly Disagree.

CONTACTS AND LOCATIONS:
Overall Officials: Zoe Diana Draelos, M.D., Principal Investigator — Dermatology Consulting Services, High Point NC
Locations (1):
- Dermatology Consulting Services, PLLC, High Point, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
Johnson & Johnson Consumer Inc. has an agreement with the Yale Open Data Access (YODA) Project to serve as the independent review panel for evaluation of requests for clinical study reports and participant level data from investigators and physicians for scientific research that will advance medical knowledge and public health. Requests for access to the study data can be submitted through the YODA Project site at http://yoda.yale.edu.
URL: http://yoda.yale.edu

REFERENCES:
- [Background] Rajka G, Langeland T. Grading of the severity of atopic dermatitis. Acta Derm Venereol Suppl (Stockh). 1989;144:13-4. doi: 10.2340/000155551441314. PMID 2800895
- See also: Related Info — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217051&parentIdentifier=CCSSKA004706&attachmentIdentifier=9784bbe0-cf4e-4cc3-9a81-2f32fcb59939&fileName=CCSSKA004706_Clinical_Study_Report_Synopsis_FINAL.pdf&versionIdentifier=